CLINICAL TRIAL: NCT02454517
Title: PALS: Prostate Cancer Active Lifestyle Study
Brief Title: Diet and Exercise Program to Promote Weight Loss and Improve Health in Men With Low- or Low-Intermediate-Risk Prostate Cancer
Acronym: PALS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to insufficient funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jonathan Wright, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 9369; NCI-2015-00686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1001233 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA184075 (NIH)
Record Dates: First submitted 2015-05-22; First posted 2015-05-27 (Estimated); Results first posted 2022-12-16 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Prostate Adenocarcinoma; Stage I Prostate Cancer AJCC V7; Stage IIA Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (diet and exercise lifestyle intervention) (Experimental): The goals of the diet and exercise lifestyle intervention is for patients to lose 7% total body weight. Patients meet with a nutritionist 11 times during the first 6 months to receive the structured diet and exercise instruction. Participants complete exercise sessions supervised by an exercise specialist, and will wear a heart rate monitor periodically during the study.
  Interventions: Behavioral: Behavioral Dietary Intervention; Behavioral: Exercise Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (control) (Active Comparator): Patients receive an informational intervention along with a 20-30 minute individual session with a dietitian and a goal of 30 minutes of physical activity 5 days a week.
  Interventions: Other: Informational Intervention; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Undergo DPP lifestyle intervention
  Arms: Arm I (diet and exercise lifestyle intervention)
Behavioral: Exercise Intervention — Undergo DPP lifestyle intervention
  Arms: Arm I (diet and exercise lifestyle intervention)
Other: Informational Intervention — Receive oral and written guidelines and meet with dietician
  Arms: Arm II (control)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase III trial studies a diet and exercise program based on the Diabetes Prevention Program to promote weight loss and improve health in men with low-risk or low-intermediate-risk prostate cancer on active surveillance. A lifestyle intervention that promotes weight loss may influence prostate health. A combined diet and exercise program that is based on the Diabetes Prevention Program may affect markers (or "biomarkers") of prostate cancer progression. Gathering this information may help doctors understand how obesity affects prostate cancer progression and may help lead to a program that can reduce the risk of prostate cancer progression.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test whether the Diabetes Prevention Program (DPP) lifestyle intervention (versus [vs.] control) improves serum fasting glucose.

II. To test whether the DPP lifestyle intervention (vs. control) improves serum biomarkers of glucose regulation (insulin, C-peptide, insulin-like growth factor-1 [IGF-1], IGF binding protein 3 [IGF-BP3] and adiponectin).

III. To test whether the DPP lifestyle intervention decreases the levels of insulin receptor or insulin-like growth factor-1 receptor (IGF-1R) in prostate cancer (PCa) tissue epithelium on follow-up prostate biopsy.

IV. To test whether PCa patients randomized to the DPP lifestyle intervention sustain the lifestyle changes for at least 6 months after the end of the intervention period.

SECONDARY OBJECTIVES:

I. To evaluate whether the DPP lifestyle intervention improves health-related quality of life.

II. To evaluate whether the DPP lifestyle intervention effects on pathologic features of follow-up prostate biopsies.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients meet with a nutritionist 11 times during the first 6 months to receive the structured diet and exercise instruction. Participants complete exercise sessions supervised by an exercise specialist, and will wear a heart rate monitor periodically during the study.

ARM II: Patients receive oral and written information based on general U.S. dietary and physical activity guidelines along with a 20-30 minute individual session with a dietitian and a goal of 30 minutes of physical activity 5 days a week.

After completion of study, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate, clinically localized, low or low-intermediate risk disease (T1C/T2a, Gleason =< 7 [3+4], prostate-specific antigen [PSA] < 20)
* Primary treatment is active surveillance (AS) with planned annual surveillance biopsies
* Body mass index (BMI) >= 25 kg/m^2; and
* Physically able to undertake a diet and exercise program

Exclusion Criteria:

* Current, recent (< 1 year), or planning to join a weight loss program or take appetite suppressants
* Steroid hormone use (antiandrogen therapy [ADT]) within the past 12 months
* Significant cardiovascular disease precluding an exercise program, including recent (within 6 months) myocardial infarction or stroke, pulmonary edema, myocarditis, pericarditis, unstable angina, pulmonary embolism/deep venous thrombosis (PE/DVT), uncontrolled hypertension (systolic blood pressure [SBP] > 200; diastolic blood pressure [DBP] > 110), uncontrolled arrhythmia, heart failure; or
* Insulin dependent diabetes mellitus (DM) and/or metformin use
* Doctor of medicine (MD) confirmed cognitive impairment
* Current alcohol or narcotic abuse

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2016-05-19 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Diet and Exercise Lifestyle Intervention): The goals of the diet and exercise lifestyle intervention is for patients to lose 7% total body weight. Patients meet with a dietitian11 times during the first 6 months to receive the structured diet and exercise instruction. Participants complete exercise sessions supervised by an exercise specialist, and will wear a heart rate monitor periodically during the study.
  Behavioral Dietary Intervention: Undergo DPP lifestyle intervention
  Exercise Intervention: Undergo DPP lifestyle intervention
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
- Arm II (Control): Patients receive an informational intervention along with a 20-30 minute individual session with a dietitian and a goal of 30 minutes of physical activity 5 days a week.
  Informational Intervention: Receive oral and written guidelines and meet with dietitian.
  Laboratory Biomarker Analysis: Correlative studies
  Quality-of-Life Assessment: Ancillary studies
  Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Started | 58 | 59
Completed | 50 | 50
Not Completed | 8 | 9
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 4 | 7
Not completed — Discontinued Active surveillance and underwent treatment | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control) | Total
Number analyzed (Participants) | 58 | 59 | 117
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 35 | 36 | 71
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66.6 [61.7 to 71.2] | 67.0 [61.8 to 69.9] | 66.6 [61.7 to 70.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 59 | 117
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 2 | 7
  White | 48 | 51 | 99
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 117
Glucose [Mean (Standard Deviation); unit: mg/dL] — Fasting Glucose
  mg/dL | 73.5 (19.1) | 76.0 (24.3) | 74.8 (21.8)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Glucose at 6 Months
Description: Mean and standard deviation of change from baseline.
Time Frame: Baseline to 6 months
Population: Participants that completed the 6 month visit
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Arm I (Diet and Exercise Lifestyle Intervention): Intervention based on the Diabetes Prevention Program for weight loss. Patients meet with a dietitian11 times during the first 6 months to receive the structured diet and exercise instruction. Participants complete exercise sessions supervised by an exercise specialist, and will wear a heart rate monitor periodically during the study.
- Arm II (Control): General guidance on weight loss, healthy diet and physical activity provided in a single session (20 - 30 minutes).
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 50 | 50
mg/dL | -3.65 (21) | 4.5 (47)

2. Primary Outcome: Change From Baseline in Fasting C-peptide, IGF-1, IGF-BP3, and Adiponectin at 6 Months
Description: Mean and standard deviation of change from baseline.
Time Frame: Baseline to 6 months
Population: Participants who completed the 6 month study visit
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 50 | 50
ng/ml
  C-peptide (ng/mL) | -0.55 (0.72) | 0.06 (0.65)
  IGF-BP3 (ng/mL) | -363 (818) | -297 (881)
  IGF-1 (ng/mL) | 6.2 (54) | -4.7 (51)
  Adiponectin (ng/mL) | 696 (3124) | 4.2 (1652)

3. Primary Outcome: Change in Expression of Insulin Receptor (IR), IGF-1R, and Protein Kinase B (AKT) on Prostate Cancer Epithelial Cells
Description: Mean and standard deviation of change from baseline.
Time Frame: Baseline (6 months prior to randomization) to follow-up surveillance biopsy (6 months post-randomization)
Population: Data were not collected due to lack of funding.
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Weight at 12 Months
Description: Mean and standard deviation of weight at 12 months
Time Frame: 12 months (6 months after active intervention)
Population: Participants who completed the month 12 study visit
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 36 | 42
kilograms | 90.0 (14.3) | 99.2 (20.1)

5. Primary Outcome: Change From Baseline in Fasting Insulin at 6 Months
Description: Mean and standard deviation of change from baseline.
Time Frame: Baseline to 6 months
Population: Participants who completed the 6 month study visit
Measure: Mean (Standard Deviation); unit: mUI/L
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 50 | 50
mUI/L | -2.3 (4.9) | -0.19 (4.6)

6. Secondary Outcome: Health Related Quality of Life (HRQOL) at 6 Months
Description: Mean and standard deviation of Quality of Life measures at 6 months.
Time Frame: 6 months
Population: Participants who completed the 6 month study visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
Number analyzed (Participants) | 50 | 49
score on a scale
  Overall Anxiety (MAX-PC); range 0-54, higher score indicates more anxiety | 16.9 (7.5) | 16.6 (6.3)
  Urinary Quality of Life (EPIC-26); range 0-100, higher score indicates better urinary QOL: number analyzed (Participants) | 49 | 49
  Urinary Quality of Life (EPIC-26); range 0-100, higher score indicates better urinary QOL | 88.1 (11.6) | 82.9 (12.7)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Arm I (Diet and Exercise Lifestyle Intervention) | Arm II (Control)
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59
Other Adverse Events (participants affected / at risk) | 17/58 | 6/59
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Diet and Exercise Lifestyle Intervention) (N=58) | Arm II (Control) (N=59)
Arthralgia (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) — Pain in joint
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Transurethral resection of the prostate (Surgical and medical procedures) | 1 (1) | 0 (0)
Rectal hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — post prostate biopsy
Cystitis, non-infective (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) — post prostate biopsy
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Rib
Shin splints (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) — Asymptomatic, discovered on ECG
Conduction disorder (Cardiac disorders) | 0 (0) | 1 (1) — Right bundle branch block; symptomatic, discovered on ECG
Premature Ventricular Complex (Cardiac disorders) | 0 (0) | 1 (1) — Asymptomatic, discovered on ECG
Atrioventricular block, 2nd degree (Cardiac disorders) | 1 (1) | 0 (0) — Asymptomatic, discovered on ECG
Acute arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) — Asymptomatic, discovered on ECG

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-20): https://cdn.clinicaltrials.gov/large-docs/17/NCT02454517/Prot_SAP_000.pdf